CLINICAL TRIAL: NCT06658860
Title: Dimensional Changes of Alveolar Ridge After Tooth Extraction Using the Socket Shield Technique Without Immediate Implant Placement.
Brief Title: Alveolar Ridge Changes Post Tooth Extraction With Socket Shield Without Immediate Implant Placement"
Acronym: CBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soaad Tolba Mohammed Tolba Badawi (Other)
Responsible Party: Sponsor-Investigator, Soaad Tolba Mohammed Tolba Badawi, Lecturer of Oral and maxillofacial Surgery, Faculty of dentistry, Mansoura university., Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A27030123
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Alveolar Ridge Resorption After Extraction
Keywords: Tooth Extraction; Modified Socket Shield Technique

STUDY DESIGN:
Intervention Model Description: This study followed a parallel-group design. Participants were randomly assigned to two groups: one received the modified socket shield technique and the other received conventional extraction without the socket shield. Both groups were monitored after 6 months to compare alveolar ridge preservation outcomes, with delayed implant placement performed in both groups at 6 months after tooth extraction.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Socket Shield Technique (Experimental): Participants in this group underwent partial tooth extraction using the modified socket shield technique to preserve the alveolar ridge for delayed implant placement. CBCT scans were used to evaluate ridge preservation over time.
  Interventions: Procedure: Modified Socket Shield Technique
- Conventional Tooth Extraction (Active Comparator): Participants in this group underwent conventional tooth extraction without the socket shield technique. The alveolar ridge was evaluated using CBCT over the same period as the experimental group for comparison.
  Interventions: Procedure: Conventional Tooth Extraction

INTERVENTIONS:
Procedure: Modified Socket Shield Technique — The modified socket shield technique involves partial retention of the buccal aspect of the tooth root during extraction to preserve the surrounding alveolar bone and soft tissue. This technique is used to optimize the condition for delayed implant placement by preventing resorption of the alveolar ridge.
  Arms: Modified Socket Shield Technique
Procedure: Conventional Tooth Extraction — Conventional tooth extraction involves the complete removal of the tooth without the use of the socket shield technique. This arm served as the control group, with alveolar ridge changes observed and compared with those in the experimental arm over time.
  Arms: Conventional Tooth Extraction

SUMMARY:
This study aimed to evaluate the dimensional changes in the alveolar ridge after tooth extraction using the socket shield technique without immediate implant placement. The changes using CBCT were assessed, focusing on the preservation of the ridge for delayed implant placement. This research could help improve dental implant outcomes by preserving bone and soft tissue structures."

DETAILED DESCRIPTION:
"In this clinical trial, the dimensional changes in the alveolar ridge following tooth extraction were investigated using the socket shield technique. The socket shield technique involved partial retention of the root structure to preserve the surrounding bone and soft tissues. No immediate implant placement was performed, and the ridge changes were assessed at multiple time points through CBCT scans. The study included a specified sample size, and participants underwent a follow-up of 6 months after socket shield preparation. This research aimed to provide insights into how well the socket shield technique preserves ridge dimensions over time, potentially optimizing future implant stability."

ELIGIBILITY:
Inclusion Criteria:

* Non-restorable teeth in the esthetic region.
* The buccal periodontal tissues were intact.
* Maintaining oral hygiene.

Exclusion Criteria:

* The usual limitations for oral surgery.
* Tooth having a vertical fracture of the root on the facial aspect.
* Tooth having horizontal fracture of the root extending below the level of the bone.
* Caries on the root segment to be maintained.
* Mobility of the tooth.
* Bruxism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Alveolar Ridge Width Changes | 6 months post-extraction
  This outcome measure assesses changes in the alveolar ridge width following tooth extraction using either the modified socket shield technique or conventional extraction. Measurements were obtained through CBCT imaging at baseline and 6 months post-extraction. Unit of Measure: Millimeters (mm)
Bone Plate Height Changes | 6 months post-extraction
  This outcome measure assesses changes in the bone plate height following tooth extraction using either the modified socket shield technique or conventional extraction. Measurements were obtained through CBCT imaging at baseline and 6 months post-extraction. Unit of Measure: Millimeters (mm)

SECONDARY OUTCOMES:
Primary Implant Stability | At the time of implant placement, typically 6 months post-extraction.
  This outcome measure assessed the primary stability of dental implants placed after using either the socket shield technique or conventional extraction. Implant stability was evaluated using resonance frequency analysis (RFA) at the time of implant placement."

CONTACTS AND LOCATIONS:
Overall Officials: Soaad T Badawi, Lecturer, Oral Surgery, MU, Principal Investigator — Faculty of dentistry, Mansoura university
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to privacy concerns and the confidential nature of patient data. Additionally, the current study protocol does not include provisions for external data sharing."

REFERENCES:
- [Background] de Oliveira GB, Rebello IMC, Montanha Andrade K, Araujo NS, Dos Santos JN, Cury PR. Evaluation of alveolar process resorption after tooth extraction using the socket shield technique without immediate installation of implants: a randomised controlled clinical trial. Br J Oral Maxillofac Surg. 2021 Dec;59(10):1227-1232. doi: 10.1016/j.bjoms.2021.04.001. Epub 2021 Apr 8. PMID 34256958